CLINICAL TRIAL: NCT04782362
Title: Validity and Reliability of the Turkish Version of the Pectus Carinatum Body Image Quality of Life Questionnaire for Patients With Pectus Carinatum
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assistant Professor, Acibadem University
Other Study IDs: 2020-19/11
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Pectus Carinatum; Quality of Life; Body Image; Brace
MeSH Terms: conditions — Pectus Carinatum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Brace Treatment — Body image and quality of life of individuals who have used brace will be evaluated

SUMMARY:
In children with severe pectus carinatum, a significant loss of self-esteem, impairment in social behavior due to a decrease in quality of life associated with physical appearance and mental health has been reported. However, a questionnaire measuring these problems specific to this disease is not available in Turkish. Therefore, in our study, we aimed to investigate the validity and reliability of the Pectus Carinatum Body Image Quality of Life Questionnaire (PeCBI-QOL) in patients with Pectus Carinatum.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with Pectus Carinatum by a doctor (2 cm above the protrusion level)
2. Between the ages of 10-18,
3. Having dissatisfaction with this defect

Exclusion Criteria:

1. Having severe scoliosis (Cobb angle over 20 degrees)
2. Having chronic systemic disease
3. Having a serious psychiatric illness
4. Having complex mixed type pectus deformity

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Pectus Carinatum
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Pectus Carinatum Body Image Quality of Life Questionnaire | 15-21 days
  A questionnaire (Pectus Carinatum Body Image Quality of Life Questionnaire, PeCBI-QOL) was developed by Paulson et al. to be applied in the follow-up of Pectus Carinatum patients. The questionnaire includes 18 items for patients and 15 items for their families. The questionnaire has no validity and reliability in Turkish.

SECONDARY OUTCOMES:
The Pectus Excavatum Evaluation Questionnaire | 15-21 days
  The Pectus Excavatum Evaluation Questionnaire (PEEQ) was developed and validated by Lawson et al to measure the physical and psychosocial quality-of-life changes after surgical repair of pectus excavatum. Each of the 17 items in the PEEQ is in a Likert scale format, where low scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Pectus Carinatum — https://www.nlm.nih.gov/